CLINICAL TRIAL: NCT03971149
Title: Examining the Feasibility of EMPOWER - A Personalized Adherence Enhancement Intervention for Older Post-discharge Heart Failure Patients
Brief Title: EMPOWER Study, a Personalized Home Care Intervention for Older Heart Failure Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We came across unexpected difficulty with recruitment.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jinjiao Wang, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RSRB00003400
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavorial intervention (Experimental)
  Interventions: Behavioral: EMPOWER

INTERVENTIONS:
Behavioral: EMPOWER — EMPOWER includes 4 weekly home visit and 4 follow up booster phone calls every other week for the following 8 weeks. The trained nurse interventionist will address identified adherence barriers related to knowledge deficits about heart failure and its treatment including psycho-social barriers and logistic barriers with their primary care physician if necessary.

SUMMARY:
The purpose of this study is to see how investigators may best improve treatment adherence and disease management for heart failure after hospital discharge. This is because the period after hospital discharge is critical to long-term recovery, overall quality of life, and prevention of future hospitalizations. In this study, a trained nurse interventionist will work with the participants to develop a personalized adherence enhancement strategy for heart failure diagnosis. The personalized adherence enhancement strategy is called EMPOWER.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate/severe heart failure at hospital admission, defined by ICD codes (ICD-9 428 or ICD-10 150), New York Heart Association class III/IV, and left ventricular ejection fraction less than or equal to 40% (i.e., echocardiography)
* discharge from heart failure-led hospitalization to home health care in approximately the previous week
* intact or mildly impaired cognitive function (Montreal Cognitive Assessment eligibility scores greater than or equal to 18)
* primary residence in four counties within 30 minutes distance to the University of Rochester

Exclusion Criteria:

* end-of-life prognosis in the following 6 months that make it difficult to examine the changes in heart failure outcomes
* currently receiving hospice care
* conditions that impact the receipt of the intervention such as active suicidal ideation that is identified at baseline using the Geriatric Depression Scale and the Geriatric Suicide Ideation Scale
* being non-English speaking
* having serious visual and or hearing impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in medication adherence | week 1 to week 4
  Adherence will be calculated either by manual pill counting or by the Medication Event Monitoring System, a microelectronic monitoring device on the cap of medication containers.
Mean change in medication adherence | week 1 to 3 months
  Adherence will be calculated either by manual pill counting or by the Medication Event Monitoring System, a microelectronic monitoring device on the cap of medication containers.
mean change in adherence to low-sodium diet | week 1 to week 4
  Adherence to low sodium diet will be assessed by the Dietary Sodium Restriction Questionnaire (DSRQ). The DSRQ is composed of 3 subscales: 1) attitude toward the behavior, 2) subjective norm, and 3) perceived behavioral control.
  Attitude. There are 6 items in the Attitude subscale. The scores on this subscale ranged from 6 to 30, where a higher score indicates correct attitudes (better knowledge) about following a low-sodium diet.
  Subjective norm. There are 3 items in the Subjective Norm subscale. The scores on this subscale ranged from 3 to 15, where a higher score indicates heavier influence of subjective norm of social contacts on one's adherence to low-sodium diet.
  Perceived behavioral control. There are 7 items in the Perceived Behavioral Control subscale. The scores on this subscale ranged from 7 to 35, a higher score indicates a higher likelihood for each item to be a barrier in adherence to low-sodium diet.
mean change in adherence to low-sodium diet | week 1 to 3 months
  Adherence to low sodium diet will be assessed by the Dietary Sodium Restriction Questionnaire (DSRQ). The DSRQ is composed of 3 subscales: 1) attitude toward the behavior, 2) subjective norm, and 3) perceived behavioral control.
  Attitude. There are 6 items in the Attitude subscale. The scores on this subscale ranged from 6 to 30, where a higher score indicates correct attitudes (better knowledge) about following a low-sodium diet.
  Subjective norm. There are 3 items in the Subjective Norm subscale. The scores on this subscale ranged from 3 to 15, where a higher score indicates heavier influence of subjective norm of social contacts on one's adherence to low-sodium diet.
  Perceived behavioral control. There are 7 items in the Perceived Behavioral Control subscale. The scores on this subscale ranged from 7 to 35, a higher score indicates a higher likelihood for each item to be a barrier in adherence to low-sodium diet.

CONTACTS AND LOCATIONS:
Overall Officials: Jinjiao Wang, PhD, RN, Principal Investigator — University of Rochester
Locations (1):
- UR Medicine Home Care, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No